CLINICAL TRIAL: NCT06425783
Title: Warmed Blood Transfusion in Premature Babies Less Than 34 Weeks of Gestational Age: a Randomized Controlled Trial
Brief Title: Warmed Blood Transfusion in Premature Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Sibel Sevuk Ozumut, pediatric clinic chief assistant, MD, Goztepe Prof Dr Suleyman Yalcın City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SYNEO-03
Record Dates: First submitted 2024-05-08; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Transfusion Related Complication; Premature
Keywords: premature infants; warmed blood transfusion; hypothermia; hemolysis
MeSH Terms: conditions — Premature Birth; Hypothermia; Hemolysis

STUDY DESIGN:
Intervention Model Description: randomized controlled, parallel group. A single center
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Transfusion (No Intervention): It was planned to transfuse the blood at +4C temperature brought from the blood bank center in 3 hours. At the end of the standard transfusion period of 3 hours, all babies will be routinely checked for blood gases, HTC and K.
- Blood transfusıon (Experimental): Blood will be warmed before transfusion. At the end of the standard transfusion period of 3 hours, all babies will be routinely checked for blood gases, HTC and K.
  Interventions: Procedure: Warmed Blood Transfusion

INTERVENTIONS:
Procedure: Warmed Blood Transfusion — The erythrocyte suspension will be heated between 34-36 C⁰, which is the determined physiological temperature.
  Before giving it to the baby, 2 ml of blood will be taken through a triple tap and its hematocrit and K value (blood gas) will be checked. It will be given to the baby after the temperature is checked with a body fluid thermometer and determined to be within the appropriate range and if hemolysis is not observed.
  At the end of the standard transfusion period of 3 hours, all babies will be routinely checked for blood gases, HTC and K.
  Arms: Blood transfusıon

SUMMARY:
Premature babies have to deal with many problems from the moment they are born due to the immature of their organs. Their clinical condition is unstable, especially in the first few weeks, and they are greatly affected by environmental factors. During this period, blood transfusion may be needed for many reasons such as intraventricular hemorrhage and necrotizing enterocolitis. In addition, multiple blood draws to evaluate irregular metabolic, hematological and biochemical findings result in anemia and the need for blood transfusion. There are many algorithms regarding blood transfusion indications and transfusion limits in premature babies. However, there are no strict rules regarding the application of warming before blood transfusion, but it is recommended by some guidelines. Especially in unstable babies such as advanced premature babies, it is recommended to give blood by heating it at physiological temperature to avoid important complications such as hypothermia, coagulopathy and rhythm disturbances. Premature babies, whose hemodynamic and metabolic balance is very sensitive, may go into hypothermia when blood and products stored at +4C⁰ are given without heating. In routine practice, blood transfusion is performed without heating. The concern here is that hemolysis may develop by heating the blood. Studies have shown that hemolysis occurs when blood is heated above 46C⁰. In this study, physiological heating is planned. In vitro neonatal experimental modeling has shown that there is no hemolysis with physiological heating.

The aim of the researchers is; While protecting fragile, extremely premature babies from the complications of cold transfusion, the aim is to compare the transfusion groups with and without physiological heating in terms of hemolysis, metabolic balance and cerebral tissue oxygenation.

DETAILED DESCRIPTION:
This trial is planned to be randomized and controlled. Erythrocyte transfusion (ET) will be applied to premature babies born below the 34th gestational week, based on the limit values specified by TND, during Level 3 routine intensive care treatment and follow-up. They will be divided into two groups of 20 babies each: control and study groups. The control group will receive erythrocyte transfusion without heating, which is routinely applied. Heated ET will be performed on the study group by physiological warming between 34-36C⁰.

Procedures to be applied for the working group:

1. ET requirement will be determined in line with the TND guide. It will be transfused at a standard dose of 20 ml/kg. Before ET is performed, blood gas and HTC, K and blood temperature before entering the heater will be measured and recorded.
2. The erythrocyte suspension will be heated between 34-36 C⁰, which is the determined physiological temperature.
3. Before giving it to the baby, 2 ml of blood will be taken through a triple tap and its hematocrit and K value (blood gas) will be checked. It will be given to the baby after the temperature is checked with a body fluid thermometer and determined to be within the appropriate range and if hemolysis is not observed.
4. At the end of the standard transfusion period of 3 hours, all babies will be routinely checked for blood gases, HTC and K.

As standard for all babies during transfusion; Heart rate, blood pressure, saturation and body temperatures will be monitored.

It was planned to investigate whether there was a difference in terms of hypothermia and hemolysis between the groups with and without Physiological Heating. It will be examined whether heated blood has an effect on cerebral tissue perfusion by NIRS monitoring

ELIGIBILITY:
Inclusion Criteria:

* Premature babies less than 34 weeks of gestation Babies requiring ES transfusions while receiving treatment in the NICU

Exclusion Criteria:

* babies with severe congenital anomalies

Ages: 1 Hour to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Effect of heated blood transfusion on body temperature in premature babies | 6 hours
  The baby's body temperature will be measured and recorded before, during and after heated and unheated blood transfusions. It will be determined whether transfusion of unwarmed blood causes lower body temperature.
Effects of warming blood in blood transfusion on cerebral tissue oxygenation | 8 hours
  Cerebral tissue oxygenation will be measured with Near infrared spectroscopy (NIRS) monitoring in both transfusion applications. The data recorded on the NIRS device will be transferred to the computer and compared. The effect of warming the blood on cerebral tissue oxygenation will be demonstrated.
Effect of heated and unheated blood transfusion on hematocrit level | 8 hours
  After the heated and unheated blood transfusion ends, the hematocrit levels of the babies will be compared to determine which model is more effective.

SECONDARY OUTCOMES:
Effect of warming blood on potassium level | 6 hours
  After the blood is brought to physiological body temperature, a sample will be taken before giving it to the baby. The presence of hemolysis will be evaluated by measuring the potassium level in blood heated at 34-36 C. At the end of the blood transfusion, potassium will be measured in the blood taken from the baby.
Effect of warming blood on LDH level | 6 hours
  After blood transfusion, LDH will be measured by taking blood samples from the babies in both groups. A measurement of LDH above 700 will be defined as hemolysis.
Effect of heated blood on blood lactate level | 8 hours
  At the end of heated and unheated blood transfusion, blood gas and blood lactate levels will be measured. It will be compared which transfusion application increases the lactate level more.

CONTACTS AND LOCATIONS:
Overall Officials: Fahri Ovalı, Prof, Study Chair — Istanbul Medeniyet University
Locations (1):
- Goztepe Prof Dr. Suleyman Yalcın City Hospital, Istanbul, N/A (n/a), Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey SM, Mally PV. Near-Infrared Spectroscopy to Guide and Understand Effects of Red Blood Cell Transfusion. Clin Perinatol. 2023 Dec;50(4):895-910. doi: 10.1016/j.clp.2023.07.006. Epub 2023 Aug 17. PMID 37866855
- [Result] Poder TG, Nonkani WG, Tsakeu Leponkouo E. Blood Warming and Hemolysis: A Systematic Review With Meta-Analysis. Transfus Med Rev. 2015 Jul;29(3):172-80. doi: 10.1016/j.tmrv.2015.03.002. Epub 2015 Mar 24. PMID 25840802
- [Result] Hulse W, Bahr TM, Fredrickson L, Canfield CM, Friddle K, Pysher TJ, Ilstrup SJ, Ohls RK, Christensen RD. Warming blood products for transfusion to neonates: In vitro assessments. Transfusion. 2020 Sep;60(9):1924-1928. doi: 10.1111/trf.16007. Epub 2020 Aug 10. PMID 32776545
- [Result] Dani C, Pratesi S, Fontanelli G, Barp J, Bertini G. Blood transfusions increase cerebral, splanchnic, and renal oxygenation in anemic preterm infants. Transfusion. 2010 Jun;50(6):1220-6. doi: 10.1111/j.1537-2995.2009.02575.x. Epub 2010 Jan 22. PMID 20113454